CLINICAL TRIAL: NCT05309772
Title: Randomised Controlled Multicentre Trial on the Clinical Impact of the Basophil Activation Test and the Mast Cell Activation Test as Food Allergy Biomarkers in Children and Young People
Brief Title: The Clinical Impact of the Basophil Activation Test to Diagnose Food Allergy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: King's College London (Other)
Collaborators: Sandwell & West Birmingham Hospitals NHS Trust (Other); Cambridge University Hospitals NHS Foundation Trust (Other); NHS Lothian (Other Government); University Hospitals, Leicester (Other); Guy's and St Thomas' NHS Foundation Trust (Other); University College London Hospitals (Other); King's College Hospital NHS Trust (Other); Manchester University NHS Foundation Trust (Other Government); Newcastle-upon-Tyne Hospitals NHS Trust (Other); Sheffield Children's NHS Foundation Trust (Other); University Hospital Southampton NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: IRAS 299511
Record Dates: First submitted 2021-09-07; First posted 2022-04-04 (Actual); Last update posted 2023-09-06 (Actual); Status verified 2023-03

CONDITIONS: Food Allergy; Food Allergy in Infants; Food Allergy in Children; Food Allergen Sensitisation; Milk Allergy; Egg Allergy; Nut Allergy
Keywords: Food allergy; Milk allergy; Egg allergy; Nut allergy; Basophil activation test; Mast cell activation test; Diagnosis; Specific IgE; Skin prick test; Oral food challenge
MeSH Terms: conditions — Food Hypersensitivity; Milk Hypersensitivity; Egg Hypersensitivity; Nut Hypersensitivity; Disease | interventions — Basophil Degranulation Test

STUDY DESIGN:
Intervention Model Description: Patients will be randomised using a 4:5 allocation between standard-of-care/biomarker arms. Stratified randomisation will be adopted according to recruiting centre, using a web-based allocation system.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Biomarker arm (Experimental): All participants will have blood taken to test for BAT/MAT. Participants with a positive BAT/MAT will dispense from oral food challenge (OFC).
  Participants with negative or inconclusive BAT/MAT will undergo OFC.
  Interventions: Diagnostic Test: Basophil activation test (BAT); Diagnostic Test: Oral food challenge (OFC)
- Standard-of-care arm (Active Comparator): All participants in the standard-of-care arm will have blood taken to test for BAT/MAT. Regardless of the result of BAT/MAT, all participants in this arm will undergo an oral food challenge, as per the current standard-of-care.
  Interventions: Diagnostic Test: Basophil activation test (BAT); Diagnostic Test: Oral food challenge (OFC)

INTERVENTIONS:
Diagnostic Test: Basophil activation test (BAT) — Basophils and mast cells are the key drivers of food allergic reactions and anaphylaxis to foods. The study team have developed new tests that measure the reaction of mast cells and basophils by flow cytometry following stimulation with allergen, the BAT and the MAT:
  • BAT uses fresh whole blood from patients added to allergen and antibodies in a test tube. The tube containing the allergic cells are then analysed one by one to estimate how many and how much express activation markers on their surface, CD63 and CD203c.
  MAT uses a human mast cell line (LAD2 cells) which are human mast cells grown in the laboratory to which patients' plasma is added in order to mimic the patients' own mast cells. Sensitised LAD2 cells are then stimulated with allergen or controls and analysed by flow cytometry to assess the expression of the activation marker CD63 on the cell surface, similar to what happens in the BAT. Results of MAT will be considered only in cases of non-responding basophils.
  Other Names: Mast cell activation test (MAT)
Diagnostic Test: Oral food challenge (OFC) — Consumption of the food suspected of causing an allergic reaction in a medically supervised environment, starting with small amounts and progressively increasing the dose at regular intervals up to a cumulative dose corresponding to an age-appropriate portion of the food.

SUMMARY:
The BAT Impact study is a prospective multicentre study in the UK using a biomarker-led study design to compare the incidence of adverse events (defined as allergic reactions during oral food challenges) in a randomized-controlled trial. Patients will either follow the standard-of-care (i.e. an oral food challenge in case of equivocal SPT/sIgE) or follow a basophil activation test (BAT)/mast cell activation test (MAT)-based strategy, i.e. patients with a positive BAT or MAT are dispensed of an oral food challenge (OFC) and patients with a negative BAT/MAT undergo an OFC.

DETAILED DESCRIPTION:
Children aged 6 months to 15 years requiring an oral food challenge to one of the study foods (milk, egg, peanut, sesame or cashew nut) will be invited to participate in the study.

Eleven centres across the UK will be recruiting participants and perforning clinical procedures, such as skin prick testing and oral food challenges (OFC), as per standard clinical care.

Participants will be randomised 4:5 to either have the standard-of-care, i.e. oral food challenge to the suspected food, or take BAT (MAT if BAT inconclusive) into account to decide whether or not OFC will be required: if BAT/MAT is positive, food allergy will be confirmed without doing OFC; if BAT/MAT is negative, participants in the biomarker arm will undergo OFC.

The primary outcome is the proportion of positive OFC in the biomarker arm compared with the standard-of-care arm.

Secondary outcomes are: number of OFC, quality of life, anxiety and costs associated with the diagnostic work-up.

ELIGIBILITY:
Inclusion Criteria:

* Children and young people aged 6 months to 15 years
* Suspected allergy to one of the study foods (peanut, cow's milk, egg, cashew, sesame) - defined as:

  * history of clinical reaction or
  * evidence of IgE sensitisation (SPT>0mm and/or specific IgE>=0.10 KU/L) to the respective food or
  * reassessment for possible resolution of allergy to the specific food following previous diagnosis of food allergy
* Need for an oral food challengeOFC to the study food
* Oral food challengeOFC to reach amount of food protein in a typical portion size for child's age
* Consent from adults with parental responsibility and assent from children and young people in an age appropriate form.

Exclusion Criteria:

* Clinically significant chronic illness other than atopic diseases;
* Previous history of severe life-threatening reaction to the suspected food with documented decrease in oxygen saturation (<90%), hypotension (≥20% reduction in systolic blood pressure) and/or admission to intensive care;
* Unwillingness to comply with study procedures, namely to undergo a diagnostic food challenge;
* Contra-indication for diagnostic food challenge, namely:

  * Uncontrolled atopic diseases (e.g. eczema, asthma, rhinitis);
  * Chronic medical conditions that pose significant risk in the event of anaphylaxis or treatment of anaphylaxis (e.g. cardiac disease, severe lung disease, pregnancy, mastocytosis);
  * Inability to discontinue medications that might interfere with assessment or safety (e.g. antihistamines, β-agonists, β-blockers, NSAIDs, ACE inhibitor, antacids);
  * Recent (within 7-14 days) treatment with systemic steroids or prolonged high-dose systemic steroids or immunosuppressants;
* Undergoing treatment with omalizumab, food or inhalant allergen immunotherapy or other systemic immunomodulatory treatment;
* Inability to stop anti-histamines prior to SPT or OFC.

Ages: 6 Months to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 398 (Estimated)
Dates: Start 2023-01-13 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
The proportion of positive oral food challenges in the biomarker arm (BAT ± MAT) compared to the standard-of-care arm | Up to 1 year
  Comparison of the ratio of positive oral food challenges in the biomarker arm compared to the standard-of-care arm.
Number of OFCs in the biomarker arm (BAT ± MAT) compared to the standard-of-care arm | Up to 1 year
  Comparison of the ratio of OFCs in the biomarker arm compared to the standard-of-care arm.

SECONDARY OUTCOMES:
The quality of life of children and parents at the start and at the end of the diagnostic work-up for food allergy as assessed by the Food Allergy Quality of Life Questionnaire. | Up to 1.5 years
  Change in quality of life score at the start and end of diagnostic work-up.
Anxiety levels of parents and children before and after diagnostic work-up as assessed by the Hospital Anxiety and Depression Questionnaire. | Up to 1.5 years
  Change in anxiety score before and after diagnostic work-up.
Anxiety levels of parents and children before and after diagnostic work-up as assessed by the State Trait Anxiety Inventory. | Up to 1.5 years
  Change in anxiety score before and after diagnostic work-up.
NHS and societal costs of food allergies during the diagnostic assessment, as measured through a bespoke form. | Up to 1.5 years
  NHS and societal costs during the six weeks before and six weeks after diagnostic work-up.

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra Santos, MD, PhD, Principal Investigator — King's College London
Locations (11):
- United Kingdom (11):
  - Sandwell and West Birmingham Hospital, Birmingham
  - Addenbrookes Hospital, Cambridge
  - Royal Hospital for Children and Young People, Edinburgh
  - Leicester Royal Infirmary, Leicester
  - Evelina London Children's Hospital, London
  - King's College Hospital, London
  - University College London Hospital, London
  - Royal Manchester Children's Hospital, Manchester
  - Great North Children's Hospital, Newcastle
  - Sheffield Children's Hospital, Sheffield
  - University Hospital Southampton, Southampton

IPD SHARING:
Plan to Share IPD: No